CLINICAL TRIAL: NCT06159179
Title: Medical Thoracoscopy for Undiagnosed Transudative and Exudative Pleural Effusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Cipto Mangunkusumo General Hospital (Other)
Collaborators: Singapore General Hospital (Other)
Responsible Party: Principal Investigator, Gurmeet Singh, MD, Head Division Respirology and Critical Illness, Internal Medicine Department, Principal Investigator, Respirology and Critical Illness Consultant, Dr Cipto Mangunkusumo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1111/UN2.RST/HKP.05.00/2022; NCT05553665 (obsolete NCT alias)
Record Dates: First submitted 2023-11-15; First posted 2023-12-06 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Medical Thoracoscopy

STUDY DESIGN:
Intervention Model Description: Hospitalized adults age 18 - 75 years old; Willing to be involved in the research; Undiagnosed transudative and exudative pleural effusion post-thoracentesis twice on right and left lung; Patients can undergo medical thoracoscopy under local anesthesia, based on ATS and BTS guideline.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- undiagnosed transudative and exudative pleural effusion (Other): Subjects with undiagnosed transudative and exudative pleural effusion will undergo medical thoracoscopy as per studies protocols.
  Interventions: Procedure: Medical thoracoscopy

INTERVENTIONS:
Procedure: Medical thoracoscopy — Medical thoracoscopy is a minimally invasive procedure to have access to pleura with combination of visual and medical instrument. The procedure is done with local and light anesthesia. Medical thoracoscopy plays role in basic diagnosis and therapeutic. A Flex-rigid thoracoscope will be inserted through the trocar cannula in the rigt or left mid axillary line of the hemithorax
  Other Names: Flex-rigid thoracoscope via trocar cannula

SUMMARY:
Indonesia is one of country that contributes the most cases of tuberculosis worldwide. Tuberculosis is the most commonly etiology of exudative pleural effusion. There have been many studies about undiagnosed exudative pleural effusion, but there are not many studies about the use of medical thoracoscopy for diagnosing transudative and exudative pleural effusion, especially on biomarkers of C-Reactive Protein (CRP), D-dimer, Adenosine Deaminase (ADA), Antinuclear Antibody (ANA), C3 C4 complements, Cancer Antigen 125 (CA-125), Xpert Mycobacterium Tuberculosis (Xpert MTB), Lupus Erythematosus cell (LE cell), cytology (effusion and smear) and histopathology. Information gained from those biomarkers via thoracenthesis and medical troracoscopy, etiology of exudative and transudative pleural effusion can be detected earlier and clearly, especially etiology of infection, autoimmune, and malignancy that further can be used to reduce patients' hospitalization period, mortality, and to develop the new therapeutic agents.

DETAILED DESCRIPTION:
Medical thoracoscopy is a minimally invasive procedure to access pleura with combination of visual and medical instrument. The procedure is performed under local anesthesia and conscious sedation. Medical thoracoscopy plays role in basic diagnotic and therapeutic. The most common indication on basic diagnostic is on pleural effusion case that has primary target to get specific diagnosis when the etiology of pleural effusion is unknown. Pleural effusion is fluid accumulation inside the pleura for about 15-20 ml. Primary aim of pleural effusion diagnosis is to differentiate exudative and transudative effusions based on Light Criteria. Most of time thoracentesis cannot give etiology of exudative and transudative pleural effusion.

Researchers will evaluate subjects based on inclusion and exclusion criteria in Cipto Mangunkusumo Hospital. Furtehrmore, research subjects will be asked for informed consent. Data will be collected based on research form. Researcher will perform medical thoracoscopy to take specimen for analysing CRP, D-dimer, ADA, ANA, C3 C4 complements, Xpert MTB, LE cell, cytology (effusion and smear) and histopathology to detect the etiology of tuberculosis, malignancy or autoimmune.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized adult age 18 - 75 years old
* Willing to be involved in the research
* Undiagnosed transudative and exudative pleural effusion post-thoracentesis twice on right and left lung
* Patients can undergo medical thoracoscopy under local anesthesia, based on ATS and BTS guideline

Exclusion Criteria:

* Pregnant and breastfeeding women
* Patients in non-invasive ventilation and mechanical ventilator
* Transudative and exudative pleural effusion with etiology of chronic heart failure, chronic kidney disease, hepatocirrhosis with or without hepatic hydrothorax and hypoalbuminemia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
To analyze role of medical thoracoscopy on undiagnosed transudative and exudative pleural effusion patients | 2 weeks
  To investigate whether medical thoracoscopy has a high diagnostic yield in undiagnosed transudative and exudative pleural effusion patients

SECONDARY OUTCOMES:
To know the prevalency of undiagnosed transudative and exudative pleural effusion. | Up to 12 months
  Number of subjects with undiagnosed transudative and exudative pleural effusion will be assessed through medical thoracoscopy
To know the etiology of infection, autoimmune and malignancy on undiagnosed transudative and exudative pleural effusion | 2 weeks
  Number of subjects with undiagnosed transudative and exudative pleural effusion will be classified for etiology of infection, autoimmune and malignancy at 2 weeks
To analyze biomarkers from blood (CRP, D-dimer, ANA, C3 C4 complements, CA-125) , , cytology (effusion and smear) and histopathology on undiagnoses transudative and exudative pleural effusion | Up to 12 months
  Results of CRP, D-dimer, ANA, C3 C4 complements, CA-125 from blood samples from subjects with undiagnosed transudative and exudative pleural effusion will be known at 12 months
To analyze biomarkers from pleural effusion (ADA, Xpert MTB, LE cell) | Up to 12 months
  Results of ADA, Xpert MTB, LE cell from pleural effusion samples from subjects with undiagnosed transudative and exudative pleural effusion will be known at 12 months
To analyze cytology (effusion and smear) and histopathology on undiagnosed transudative and exudative pleural effusion | Up to 12 months
  Results of cytology and histopathology from subjects with undiagnosed transudative and exudative pleural effusion will be known at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gurmeet Singh, MD, Phd, Principal Investigator — Dr Cipto Mangunkusumo General Hospital
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Light RW. Clinical practice. Pleural effusion. N Engl J Med. 2002 Jun 20;346(25):1971-7. doi: 10.1056/NEJMcp010731. No abstract available. PMID 12075059
- [Background] Rodriguez-Panadero F, Janssen JP, Astoul P. Thoracoscopy: general overview and place in the diagnosis and management of pleural effusion. Eur Respir J. 2006 Aug;28(2):409-22. doi: 10.1183/09031936.06.00013706. No abstract available. PMID 16880371
- [Background] Ferreiro L, Toubes ME, San Jose ME, Suarez-Antelo J, Golpe A, Valdes L. Advances in pleural effusion diagnostics. Expert Rev Respir Med. 2020 Jan;14(1):51-66. doi: 10.1080/17476348.2020.1684266. Epub 2019 Nov 5. PMID 31640432